CLINICAL TRIAL: NCT06918223
Title: Assessing Patient Satisfaction and Confidence After Use of Educational Video to Augment Surgical Consent for Thyroid Surgery
Acronym: TISCAV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20E.663; STRYKER (Other Grant/Funding Number: AHNS Endocrine Surgery Section Stryker Research Award)
Record Dates: First submitted 2025-03-18; First posted 2025-04-09 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: TISCAV (Experimental)
  Interventions: Behavioral: Thyroid Informed Surgical Consent Augmenting Video (TISCAV)
- Control: Standard Consent (Placebo Comparator)
  Interventions: Behavioral: Standard Consent

INTERVENTIONS:
Behavioral: Thyroid Informed Surgical Consent Augmenting Video (TISCAV) — Participants randomized to the intervention group will receive a surgeon-created Thyroid Informed Surgical Consent Augmenting Video (TISCAV). This 8-minute video includes animated visuals and a surgeon voiceover explaining thyroid anatomy, surgical options (lobectomy vs. total thyroidectomy), risks, benefits, and expectations. The TISCAV was designed and reviewed by an endocrine surgery team to improve patient comprehension, confidence, satisfaction, and reduce decision regret compared to standard verbal consent alone.
  Arms: Intervention: TISCAV
Behavioral: Standard Consent — Participants receiving the Standard Consent intervention will undergo the routine informed consent process for thyroid surgery provided by their surgeon. This process includes a verbal discussion covering thyroidectomy procedure details, potential risks and complications, benefits, alternatives such as active surveillance, and an opportunity to ask questions.
  Arms: Control: Standard Consent

SUMMARY:
This study looks at how a short educational video can help people better understand thyroid surgery. Patients who have thyroid nodules and need surgery will be part of the study. Some patients will get the usual information from their doctor, while others will also watch a video that explains the surgery in a simple and clear way. The study will check if the video helps patients feel more confident about their decision, lowers anxiety, and helps them remember important information about their surgery. Patients will answer surveys before surgery, after surgery, and 3 months later.

ELIGIBILITY:
Inclusion Criteria Fluent in English

* English is Primary Language
* ≥18 years old at time of consent
* Eligible for Thyroidectomy, lobectomy, isthmusectomy for any indication

Exclusion Criteria:

* History of prior thyroid surgery
* Previously consented for thyroid surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Patient knowledge score using a 10-item internally validated Thyroid Surgery Knowledge Assessment | Immediately after study enrollment (pre-consent) and immediately following the surgical consent process (post-consent)
  This outcome measures patient knowledge of thyroid surgery, including indications, procedural options, risks, and benefits. A 10-question internally developed and validated multiple-choice questionnaire will be administered before and after the informed consent process. Each correct answer is scored as 1 point, with a total score ranging from 0 to 10. Higher scores indicate greater understanding and retention of surgical information.
Decisional Conflict Score using the Decisional Conflict Scale (DCS) | Preoperatively (after the consent process and before surgery)
  This outcome measures patient uncertainty and confidence related to thyroid surgery decision-making using the validated 16-item Decisional Conflict Scale (DCS). The DCS evaluates five subdomains: uncertainty, feeling informed, values clarity, support, and perceived effectiveness of the decision. Each item is scored from 0 (strongly agree) to 4 (strongly disagree), then standardized to a total score ranging from 0 to 100. Higher scores reflect greater decisional conflict and more difficulty with making a decision.
Satisfaction with Decision Score using the Satisfaction with Decision Scale (SDS) | Immediately after consent (Preoperative), Postoperative Day 22, and Postoperative Day 100
  This outcome assesses patient satisfaction with their decision to undergo thyroid surgery using the validated 6-item Satisfaction with Decision Scale (SDS). Each item is scored from 1 (not satisfied) to 5 (very satisfied), with a total score ranging from 6 to 30. Higher scores indicate greater satisfaction with the decision-making process and outcome.
Decision Regret Score using the Decision Regret Scale (DRS) | Postoperative Day 22 and Postoperative Day 100
  This outcome evaluates postoperative regret related to undergoing thyroid surgery using the validated 5-item Decision Regret Scale (DRS). Each item is scored from 1 (strongly agree) to 5 (strongly disagree), with scores converted to a 0-100 scale. Higher scores reflect greater decision regret.
Anxiety Score using the Visual Analog Scale for Anxiety (VAS-A) | Immediately after consent (Preoperative), Postoperative Day 22, and Postoperative Day 100
  This outcome measures patients' current level of anxiety using the validated Visual Analog Scale for Anxiety (VAS-A), a single-item scale presented as a 100 mm line ranging from "calm" to "anxious." Participants place a mark on the scale reflecting their current state. The score is recorded as a number from 0 to 100, with higher scores indicating greater anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Cottrill Assistant Professor and Program Director, MD, Principal Investigator — Assistant Professor and Program Director
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated and analyzed during this study will not be publicly available due to patient confidentiality and institutional data-sharing policies. However, de-identified participant-level data (IPD) may be shared with qualified researchers upon reasonable request to the corresponding author, subject to institutional and ethical approvals. The data will be made available for research purposes related to patient comprehension, decision-making, and informed consent in surgical settings. Access will be granted following approval of a research proposal and a signed data access agreement.
Supporting Information: CSR

REFERENCES:
- [Background] Levy N, Landmann L, Stermer E, Erdreich M, Beny A, Meisels R. Does a detailed explanation prior to gastroscopy reduce the patient's anxiety? Endoscopy. 1989 Nov;21(6):263-5. doi: 10.1055/s-2007-1012965. PMID 2612430
- [Background] Kindler CH, Harms C, Amsler F, Ihde-Scholl T, Scheidegger D. The visual analog scale allows effective measurement of preoperative anxiety and detection of patients' anesthetic concerns. Anesth Analg. 2000 Mar;90(3):706-12. doi: 10.1097/00000539-200003000-00036. PMID 10702461
- [Background] Thomas T, Robinson C, Champion D, McKell M, Pell M. Prediction and assessment of the severity of post-operative pain and of satisfaction with management. Pain. 1998 Apr;75(2-3):177-85. doi: 10.1016/s0304-3959(97)00218-2. PMID 9583753
- [Background] McCleane GJ, Cooper R. The nature of pre-operative anxiety. Anaesthesia. 1990 Feb;45(2):153-5. doi: 10.1111/j.1365-2044.1990.tb14285.x. PMID 2321720
- [Background] Domar AD, Everett LL, Keller MG. Preoperative anxiety: is it a predictable entity? Anesth Analg. 1989 Dec;69(6):763-7. PMID 2589657
- [Background] D'Souza V, Blouin E, Zeitouni A, Muller K, Allison PJ. Do multimedia based information services increase knowledge and satisfaction in head and neck cancer patients? Oral Oncol. 2013 Sep;49(9):943-949. doi: 10.1016/j.oraloncology.2013.06.005. Epub 2013 Jul 16. PMID 23870712
- [Background] Hakimi AA, Standiford L, Chang E, Wong BJ. Development and Assessment of a Video-Based Intervention to Improve Rhinoplasty Informed Consent. Facial Plast Surg. 2021 Oct;37(5):585-589. doi: 10.1055/s-0041-1722912. Epub 2021 Feb 25. PMID 33634455
- [Background] Siu JM, Rotenberg BW, Franklin JH, Sowerby LJ. Multimedia in the informed consent process for endoscopic sinus surgery: A randomized control trial. Laryngoscope. 2016 Jun;126(6):1273-8. doi: 10.1002/lary.25793. Epub 2015 Nov 30. PMID 26615812
- [Background] Nehme J, El-Khani U, Chow A, Hakky S, Ahmed AR, Purkayastha S. The use of multimedia consent programs for surgical procedures: a systematic review. Surg Innov. 2013 Feb;20(1):13-23. doi: 10.1177/1553350612446352. Epub 2012 May 14. PMID 22589017
- [Background] Sudore RL, Landefeld CS, Williams BA, Barnes DE, Lindquist K, Schillinger D. Use of a modified informed consent process among vulnerable patients: a descriptive study. J Gen Intern Med. 2006 Aug;21(8):867-73. doi: 10.1111/j.1525-1497.2006.00535.x. PMID 16881949
- [Background] Burns P, Keogh I, Timon C. Informed consent: a patients' perspective. J Laryngol Otol. 2005 Jan;119(1):19-22. doi: 10.1258/0022215053222860. PMID 15807957
- [Background] Hekkenberg RJ, Irish JC, Rotstein LE, Brown DH, Gullane PJ. Informed consent in head and neck surgery: how much do patients actually remember? J Otolaryngol. 1997 Jun;26(3):155-9. PMID 9176798
- [Background] Oosthuizen JC, Burns P, Timon C. The changing face of informed surgical consent. J Laryngol Otol. 2012 Mar;126(3):236-9. doi: 10.1017/S0022215111003021. Epub 2011 Nov 4. PMID 22051081
- [Background] Kessels RP. Patients' memory for medical information. J R Soc Med. 2003 May;96(5):219-22. doi: 10.1177/014107680309600504. No abstract available. PMID 12724430
- [Background] Sherlock A, Brownie S. Patients' recollection and understanding of informed consent: a literature review. ANZ J Surg. 2014 Apr;84(4):207-10. doi: 10.1111/ans.12555. PMID 24812707
- [Background] Mulsow JJ, Feeley TM, Tierney S. Beyond consent--improving understanding in surgical patients. Am J Surg. 2012 Jan;203(1):112-20. doi: 10.1016/j.amjsurg.2010.12.010. Epub 2011 Jun 8. PMID 21641573

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-28): https://cdn.clinicaltrials.gov/large-docs/23/NCT06918223/Prot_SAP_001.pdf